CLINICAL TRIAL: NCT02321345
Title: Feasibility of Implementing Pretransplant Evaluation by the Supportive Care Team for Patients Undergoing Hematopoietic Cell Transplantation for Hematological Malignancies
Brief Title: Pretransplant Evaluation by Supportive Care Team for Patients Undergoing HCT for Hematological Malignancies
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical College of Wisconsin (Other)
Responsible Party: Principal Investigator, Wendy Peltier, MD, Medical College of Wisconsin
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 21301
Record Dates: First submitted 2014-10-18; First posted 2014-12-22 (Estimated); Last update posted 2018-02-23 (Actual); Status verified 2018-02

CONDITIONS: Malignancies, Hematologic
Keywords: Allogeneic Stem Cell Transplant; Hematological Malignancies; Palliative Care; Supportive care
MeSH Terms: conditions — Hematologic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Palliative Care Support (Experimental): Palliative care meetings will address the following issues: 1) values and meaning of life 2) greatest hopes and fears 3) communication preferences 4) proxy readiness to make decisions, and patient preferences, if the patient were to become seriously ill, and 5) symptom management strategies.
  Interventions: Other: Palliative Care Support

INTERVENTIONS:
Other: Palliative Care Support — Palliative care meetings Quality of Life Assessments

SUMMARY:
This is a feasibility study of pre-transplant involvement of a palliative care provider in the setting of HCT. Although this is primarily a feasibility pilot, the investigators will explore how patients are affected by the palliative care meetings as well as test data collection mechanisms that would be used in a future randomized clinical trial.

The investigators hypothesis is that patients will be amenable to pre-transplant involvement of the palliative care team and might welcome the chance to discuss palliative care issues separate from the primary team. Palliative care providers also have special training and experience in conducting these interactions and expertise in supportive care practices. They will be available should a patient's condition become life- threatening. This study is therefore designed primarily to evaluate the level of comfort / distress of patients when a palliative care consultation and follow-up are integrated into their care.

DETAILED DESCRIPTION:
After the patient provides written informed consent, they will be given a survey to collect baseline data. Because input may be solicited from the caregiver, consent will also be obtained from a caregiver. Participation is optional for the caregiver and a caregiver is not required for the participant to be in the study. If the caregiver does not consent to participate in the study, his/her input during meetings will not be documented in the research record. "Caregiver" may vary from patient to patient, but for the purposes of this study would be an individual who listens to the interview and responds to questions related to the patient's psychosocial history, goals and values. This information gathered from the caregiver supports the details of the consult but does not stand alone. The caregiver does not complete an evaluation of the interview but can reach out to study coordinators if the interview causes any distress.The first consultation will be scheduled with a palliative care provider, but will take place after the standard of care meeting with the social worker so that the palliative care clinician can read the social work note and not have to review the same information. Within one to seven days after the meeting with palliative care, patients will be asked to complete a 15 minute interview to provide feedback on the meeting. A brief questionnaire will also be administered to the palliative care provider who conducted the consultation, ideally immediately after the meeting. Patients will meet at least monthly with the palliative care provider while they remain at the transplant center. Patients will complete additional self-assessments at day 60+/- 7 days and 90+/- 7 days after their transplants. These surveys may be completed by mail if the patient has been discharged from the center. The medical records of participants will be reviewed to pilot items collecting data about references to the palliative care consultation and use of ACP within the first 100 days after HCT. Costs for participants will be retrieved from the inpatient and outpatient accounting systems for the first 100 days after HCT. Participants may decline to participate in any part of the study or discontinue participation at any time.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* English as primary language
* Planned allogeneic stem cell transplantation
* At least 18 years of age

Exclusion Criteria:

* Major psychiatric diagnosis that impairs cognitive functioning or is not controlled at the time of the approach, as judged by the patient's medical team.
* First transplant of a planned tandem procedure (the second transplant is eligible)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2015-02; Primary Completion 2017-10 (Actual); Study Completion 2017-10 (Actual)

PRIMARY OUTCOMES:
Study participation rates | 1 year
  The proportion of patients who consent to enroll in the study will be computed based on the number approached. Reasons for non-participation will be summarized.

SECONDARY OUTCOMES:
Completion time for palliative care consultation | up to 100 days
Level of comfort / distress attributed to individual parts of the consultation | Within 1-7 days after the initial consultation
  The post-consultation scores measuring level of comfort or distress per topic in the palliative care consultation will be summarized per item.
Completeness of follow-up data collection | 1 year after the date last patient is enrolled
  Completeness is defined by the proportion of instrument scores that can be calculated per given time point. The completeness of follow-up data collection will be calculated and reported as a proportion of successfully completed scales vs. scales attempted to be collected or completed by patients.

CONTACTS AND LOCATIONS:
Overall Officials: Wendy Peltier, MD, Principal Investigator — Medical College of Wisconsin
Locations (1):
- Froedtert Hospital and the Medical College of Wisconsin, Milwaukee, Wisconsin, United States